CLINICAL TRIAL: NCT00813852
Title: The Study of Skeletal Muscle Function in Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200612106R
Record Dates: First submitted 2008-12-21; First posted 2008-12-23 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; skeletal muscle; magnetic stimulation; magnetic resonance spectroscopy; inflammatory markers; exercise
MeSH Terms: conditions — Sleep Apnea, Obstructive; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Experimental): exercise training, CPAP, and inspiratory muscle strengthening program
  Interventions: Behavioral: exercise training, IMT

INTERVENTIONS:
Behavioral: exercise training, IMT — Each exercise session includes graded treadmill walking and resisted exercises. The graded treadmill walking exercise begins with a 5 minute warm-up period with the intensity of about 40% of maximal oxygen consumption (VO2max) follows by a 30 minutes training phase. The training intensity is set at about 70%-85% of VO2max and ends with a 5-minute cool-down period with the intensity of about 40% of VO2max. The resisted exercise program includes 20 minutes of weight training with rest after the first 5 minutes.
  Other Names: exercise

SUMMARY:
The purposes of this study includes (1)to investigate inspiratory muscles and non-inspiratory muscle function in terms of strength, endurance, and fatigability in patients with obstructive sleep apnea (OSA), (2) investigate the metabolic characteristics of peripheral muscles and biochemistry markers in patients with OSA, and (3) to detect the effect of exercise training on the measured parameters in patients with OSA.

DETAILED DESCRIPTION:
It has become increasingly recognized that skeletal muscle abnormalities are common and profound in patients with chronic inflammatory status. Based on the unique character of obstructive sleep apnea (OSA), repeated intermittent apnea and hypopnea caused by the upper airway muscles collapse during inspiration, it is logical to speculate some adaptations in skeletal muscle of patients with OSA. The purpose of the first part is to investigate the inspiratory muscle function in patients with different severity of OSA. Participants firstly underwent polysomnography assessments will be recruited. The measurements includes Epworth sleepiness scale, strength and endurance of inspiratory muscles, and fatigue test during either maximal voluntary efforts or in response to cervical magnetic stimulation (CMS) with simultaneously sEMG recordings. In addition, the exercise capacity with simultaneous sEMG recordings for diaphragm and vastus lateralis during the exercise testing will also be tested. The second part is designed to examine the metabolic characteristics of lower extremity in patients with OSA. Blood samples will be drawn and proton magnetic resonance spectroscopy is used to detect intramyocellular and extramyocellular lipid contents (IMCL and EMCL). The third part will detect the effect of exercise training on the measured parameters described as above in patients with OSA. Participants will be randomized into exercise group, inspiratory muscle training group (IMT), and CPAP group. Exercise protocol includes 30-minute aerobic exercise at the intensity of 70%-85% VO2max, and 20-minute general resistance exercise. IMT group will receive inspiratory muscle strengthening by device.

ELIGIBILITY:
Inclusion Criteria:

* ages from 40-65 years men who first underwent polysomnography at the Sleep Research Center.

Exclusion Criteria:

* Subjects who had active medical or nervous system diseases, abnormal pulmonary function, morbid obesity, diabetes managed with oral hypoglycemic agents, alcoholism (≥ 50 gm per day), or a recent infection.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
strength, endurance, fatigability, and nerve conduction velocity in response to magnetic stimulation | 4 months

SECONDARY OUTCOMES:
biochemistry markers, magnetic resonance spectroscopy | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Yueh Chien, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chien MY, Lee PL, Yu CW, Wei SY, Shih TT. Intramyocellular Lipids, Insulin Resistance, and Functional Performance in Patients with Severe Obstructive Sleep Apnea. Nat Sci Sleep. 2020 Jan 28;12:69-78. doi: 10.2147/NSS.S232554. eCollection 2020. PMID 32095087
- [Derived] Chien MY, Lee P, Tsai YF, Yang PC, Wu YT. C-reactive protein and heart rate recovery in middle-aged men with severe obstructive sleep apnea. Sleep Breath. 2012 Sep;16(3):629-37. doi: 10.1007/s11325-011-0549-2. Epub 2011 Jun 27. PMID 21706288